CLINICAL TRIAL: NCT00603655
Title: Assessment of Glycemic Load on Body Composition Among Overweight and Obese Adults During 12 Month Period
Brief Title: Effect of Glycemic Load on Body Composition
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Higher drop out than expected. Lower Statistical Power.
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Arturo Jiménez-Cruz, Universidad Autónoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UABC4268; UABC20074268
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Overweight; Obesity
Keywords: Diet; glycemic load; overweight; obesity; hyperlipidemia
MeSH Terms: conditions — Overweight; Obesity; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): This group will receive a low glycemic load
  Interventions: Other: Low glycemic load diet
- B (Active Comparator): This group will receive a high glycemic load
  Interventions: Other: High glycemic load diet

INTERVENTIONS:
Other: Low glycemic load diet — Low glycemic load diet
  Other Names: Low glycemic index
  Arms: A
Other: High glycemic load diet — High glycemic load diet
  Arms: B

SUMMARY:
The aim of this study is to compare the effects of diets with different glycemic load (GL) on body composition and biochemical markers in overweight and obese subjects during a 12-month period.

DETAILED DESCRIPTION:
Study Procedure:

The study is a randomized, experimental, parallel design conducted in a group of Mexican subjects during a 6-month period. Anthropometric and biochemical data will be determined at 0, 3, 6, 9 and 12 months.

Subjects:

Overweight or obese adults were assigned into two groups: LGL diet and HGL diet. Subjects who were pregnant or had diabetes, cancer, psychiatric disorders or physical disabilities were excluded.

Diets and Dietary Assessment:

Two diets were designed including LGL and HGL diets. GI values of each food were estimated from the tables by Foster-Powell et al. Daily GL was determined by the product of total dietary carbohydrate (grams) and GI of each food and adjusted to energetic intake using the following formulas: GI = Σ (GI of each food X proportion of total carbohydrate contributed from each food); GL= Σ (GI of each food × grams of total carbohydrate from each food)/1000 kcal.

Diets were designed according to the food habits of Mexicans living in the Tijuana area. On the first day, subjects received different menus of either LGL or HGL diets, according to the randomization. A research assistant was available by mail or by phone for questions during the 6-month period. An e-mail, as a reminder and reinforcement to maintain the diet, was sent every 2 weeks to all participants. Subjects who completed the 3-day dietary record (two weekdays and one weekend day) were included in the analysis.

Anthropometric Measurements:

Height was measured to the nearest millimeter using a portable stadiometer (model 214 Road Rod, Seca Corp., Hanover, MD). Weight was measured to the nearest 0.1 kg using an electronic scale (Bod Pod, Life Measurement Inc., Concord, CA). Subjects were dressed in light clothing and were not wearing shoes. Body mass index (BMI) was calculated using the following formula: weight (kg)/height (m2). Waist circumference (WC) was measured at the minimum circumference between the iliac crest and the rib cage. Fat mass (in kg) and total body fat percentage were measured by plethysmography with the Bod Pod. The subjects entered the Bod Pod wearing a bodysuit and Lycra hat.

Blood Analysis:

Venous blood samples were taken at 8 AM from an antecubital vein after a 12-hour overnight fast, again at baseline and at 3 months after beginning the study. Blood samples were centrifuged at 3500 × g for 3 minutes, and plasma was removed and analyzed immediately after collection. For quantitative determination of glucose in serum, the glucose oxidase procedure based on a modified Trinder method was used (SERA-PAK Plus, Bayer, Sées, France). Serum insulin levels were determined by chemiluminescent immunoassay by the IMMULITE 2000 analyzer (Diagnostic Products Corporation, Los Angeles, CA). Homeostasis model assessment (HOMA) was used to estimate insulin resistance and was computed as follows: (fasting serum insulin [μU/ml] × fasting plasma glucose [mmol/L]/22.5). Total cholesterol, HDL-cholesterol and triglycerides were measured by enzymatic methods (SERA-PAK Plus); LDL-cholesterol was calculated using the Friedwald formula: LDL (mmol/L) = total cholesterol - (TG/2.2) - HDL.

Physical Activity Assessment:

A questionnaire containing seven questions from the International Physical Activity Questionnaire (IPAQ) was used to evaluate physical activity at baseline and at 1, 3 and 6 months after study initiation.

Statistical Analysis:

Mean ± standard deviations were calculated using descriptive statistics in all variables. Anthropometric measurements were evaluated, and it was determined that they did not meet the normality test (Kolmogorov-Smirnov and Shapiro-Wilk). To test differences between groups on biochemical and anthropometric measurements, Mann-Whitney non-parametric test for independent samples was performed. For comparison of differences before, at 3 and 6 months after intervention in the same treatment group, we used Friedman non-parametric test for repeated measurements. To test differences between groups on diet intake at baseline and at the end of the study, Mann-Whitney non-parametric test for independent samples was performed.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese adults

Exclusion Criteria:

* Subjects who are pregnant or have diabetes, cancer, psychiatric disorders or physical disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of body fat percentage | 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Reduction of homeostasis model assessment (HOMA) | 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Jimenez-Cruz, MD, Principal Investigator — Universidad Autonoma de Baja California
Locations (1):
- Facultad de Medicina y Psicología, Tijuana, Estado de Baja California, Mexico